CLINICAL TRIAL: NCT03965858
Title: A Multicentre, Double-blind, Randomised, Placebo - Controlled Phase II Study to Assess Efficacy, Safety and Pharmacokinetics of Inhaled Esketamine in Subject With Treatment-resistant Depression in the Course of Major Depressive Disorder
Brief Title: Efficacy, Safety and Pharmacokinetic Study of Inhaled Esketamine in Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02KET2018
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Esketamine low dose (Experimental): Participants are to receive four doses of Esketamine DPI administered over 14-day period (on Day 1, 4, 8 and 11).
  Interventions: Drug: Esketamine DPI - low dose
- Esketamine medium dose (Experimental): Participants are to receive four doses of Esketamine DPI administered over 14-day period (on Day 1, 4, 8 and 11).
  Interventions: Drug: Esketamine DPI - medium dose
- Esketamine high dose (Experimental): Participants are to receive four doses of Esketamine DPI administered over 14-day period (on Day 1, 4, 8 and 11).
  Interventions: Drug: Esketamine DPI - high dose
- Placebo (Placebo Comparator): Participants are to receive four doses of Placebo DPI administered over 14-day period (on Day 1, 4, 8 and 11).
  Interventions: Drug: Placebo DPI

INTERVENTIONS:
Drug: Esketamine DPI - low dose — Esketamine DPI is to be administered via dry powder inhaler. Each dose correspond to low Esketamine dose.
  Arms: Esketamine low dose
Drug: Esketamine DPI - medium dose — Esketamine DPI is to be administered via dry powder inhaler. Each dose correspond to medium Esketamine dose.
  Arms: Esketamine medium dose
Drug: Esketamine DPI - high dose — Esketamine DPI is to be administered via dry powder inhaler. Each dose correspond to high Esketamine dose.
  Arms: Esketamine high dose
Drug: Placebo DPI — Placebo DPI is to be administered via dry powder inhaler.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the efficacy, safety and pharmacokinetics of inhaled Esketamine in participants with treatment-resistant depression (TRD) in the course of Major Depressive Disorder (MDD). The study is to determine the efficacy and dose response of three Esketamine doses, compared with placebo.

DETAILED DESCRIPTION:
This is a randomized, multiple dose, placebo-controlled, double-blind, multicentre study of Esketamine DPI, inhalation powder delivered via dry powder inhaler (DPI) in participants with TRD in the course of MDD. There are 3 study phases: Screening phase, a two weeks double-blind treatment phase and a 6-week follow-up phase. Participants are to be randomized in 1:1:1:1 ratio to receive placebo or one of the three doses of Esketamine DPI. Participants from each group will receive different dosing sequences, consider as a single dose, corresponding to low, medium, high Esketamine dose or placebo. Participants will undergo one cycle of treatment consisting of four doses of Esketamine DPI or placebo over 14-day period. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: female or male,
2. Age: 18 - 65 years old, inclusive, on the day of Screening,
3. Participant must meet Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) diagnostic criteria for major depressive disorder, without psychotic features, confirmed by the Mini International Neuropsychiatric Interview (MINI),
4. Participant must have in Montgomery-Asberg Depression Rating Scale (MADRS) total score of >= 25 at Screening and predose on Day 1,
5. Participant is treatment resistant, defined as having an inadequate response to at least 2 antidepressants administered for the sufficient duration and dose, both in the current episode of depression,
6. Participant must be on stable monotherapy with antidepressant drug (listed in the protocol) remain non-responsive to it and continue on non-investigational antidepressant therapy from Screening to at least the duration of the double-blind treatment phase,
7. Participant agrees to be hospitalized voluntarily for a period of 12 h before first administration and until the Day 6 of treatment phase. Hospitalization from Day 6 up to the end of treatment phase on Day 14 is up to Investigator discretion, with exception of mandatory hospitalization from 12 h before each administration until 24 h post each administration and from evening on Day 13 until the end of examinations on Day 14,
8. Participant must be medically stable on the basis of clinical laboratory tests, physical examination, vital signs, 12-lead ECG,
9. Participant agrees to blood sample collection for DNA analysis,
10. Participant of childbearing potential willing to use acceptable forms of contraception.

Exclusion Criteria:

1. Participant has a current DSM-5 diagnosis, according to MINI, of any other than MDD disorder,
2. Participant has suicidal ideation in MADRS 'suicidal thoughts' subscale score greater or equal to 2 and/or in C-SSRS score greater or equal to 4 at Screening and/or has a history of suicidal thoughts within 6 months prior to Screening and/or history of suicidal attempt within 1 year prior to Screening,
3. Participant has a history or current signs and symptoms of chronic obstructive pulmonary disease (COPD), asthma, liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, hematologic, neurologic, rheumatologic or metabolic disturbances that are uncontrolled with medication change during last three months before Screening and/or that could influence the present general health condition at the Investigator's discretion,
4. Participant has uncontrolled hypertension,
5. Upper respiratory tract and/or chest infection and/or inflammation within 2 weeks preceding the first administration and during the treatment phase,
6. Participant took part in other clinical trial within 90 days preceding the Screening,
7. Known allergy or hypersensitivity, intolerance or contraindication to Esketamine/ketamine or its derivatives and/or to any study product excipients,
8. Blood drawn within 30 days prior to inclusion to the study,
9. History of drug, alcohol, chemical, sedatives or sleeping medications abuse or dependence (except nicotine or caffeine) within 2 years prior to Screening,
10. Lifetime abuse or dependence on ketamine or phencyclidine,
11. Positive results from pregnancy test for female participants,
12. Lactation in female participants,
13. Positive drug screen (except benzodiazepines evaluation during follow-up) or alcohol breath test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score at Day 14 | Day 1 and Day 14
  The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The test consists of 10 items, each scored from 0 (symptoms not present or normal) to 6 (severe or continuous presence of the symptoms). Total score is 60. The higher MADRS total score, the more severe depression.

SECONDARY OUTCOMES:
Change from baseline in MADRS total score at each other than Day 14 timepoint | Day 1, 2, 4, 5, 8, 9, 11, 12 and week 3, 4, 5, 6, 7 and 8
  The MADRS is a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant treatment. The test consists of 10 items, each scored from 0 (symptoms not present or normal) to 6 (severe or continuous presence of the symptoms). Total score is 60. The higher MADRS total score, the more severe depression.
Number of participants with clinical response (>= 50% decrease in MADRS baseline score) | Day 1, 2, 4, 5, 8, 9, 11, 12, 14 and up to 6 weeks after the treatment phase
  Clinical response is to be defined as greater than or equal to 50 % decrease in MADRS baseline score at Day 14 and every other timepoint.
Onset of clinical response that was sustained through the end of the 2-week, double-blind, treatment phase | Day 1, 2, 4, 5, 8, 9, 11, 12, 14
Change from baseline in depression severity, measured by Hamilton Depression Rating Scale (HDRS) at every timepoint | Day 1, 2, 4, 5, 8, 9, 11, 12, 14 and week 3, 4, 5, 6, 7 and 8
  HDRS is a questionnaire used to rate the severity of depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss and somatic symptoms. HDRS consists of 17 questions with maximum 4-points scale. The higher HDRS total score, the more severe depression.
Number of participants with clinical remission (MADRS total score <= 10) | Day 1, 2, 4, 5, 8, 9, 11, 12, 14 and up to 6 weeks after the treatment phase
  Clinical remission, defined as MADRS total score less than or equal to 10.
Time to relapse | Day 14 and week 3, 4, 5, 6, 7 and 8
  Relapse assessed for responders and remitters and defined when MADRS total score in 2 consecutive assessments after Day 14 exceeds 50% MADRS baseline total score value.
Change from baseline in Clinical Global Impression - Severity (CGI-S) score at Day 14 and every other timepoint | Day 1, 2, 4, 5, 8, 9, 11, 12, 14 and week 3, 4, 5, 6, 7 and 8
  CGI-S scale is a physician-rated scale that is designed to rate the severity of the patient's illness at the time of assessment. It is a 7-point assessment where 1 = normal (not at all ill) and 7 = among the most extremely ill patients.
Change from baseline in Columbia Suicide Severity Rating Scale (C-SSRS) at Day 14 and every other timepoint | Day 1, 14 and week 5, 8
  C-SSRS is a suicide ideation rating scale created by researchers at Columbia University.
Change from baseline in the Clinician Administered Dissociative States Scale (CADSS) at each day of administration | up to 24 hours following the start of each administration
  CADSS is a scale designed to assess dissociative symptoms. CADSS consists of 23 questions with 4-points scale, where 1=normal (not at all) and 4=Extremely. The higher CADSS total score, the more severe symptoms.
Change from baseline in the Brief Psychiatric Rating Scale (BPRS) at each day of administration | up to 24 hours following the start of each administration
  BPRS is a scale designed to rate psychotomimetic effects. BPRS consists of 18 questions with 7-points scale, from 1 (not present) to 7 (extremaly severe). The higher BPRS total score, the more severe effects.
Potential withdrawal symptoms after Esketamine treatment, as measured by the 20-item Physician Withdrawal Checklist (PWC-20) | Day 0, week 3, 4 and 5
  PWC-20 is a method to assess discontinuation symptoms.
Potential Esketamine effect on cognition as measured by Montreal Cognitive Assessment (MoCA) | Day 0, week 4 and 8
  MoCA is a screening assessment for detecting cognitive impairment.
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to 8 weeks
Esketamine AUC0-24h - area under the plasma concentration - time curve from time 0 to 24 h | up to 24 hours following the start of first and fourth administration
Esketamine Cmax - maximum plasma concentration | up to 24 hours following the start of first and fourth administration
Esketamine AUC0-inf - area under the plasma concentration - time curve from time 0 to infinity | up to 24 hours following the start of first and fourth administration
Esketamine Kel - terminal elimination rate constant | up to 24 hours following the start of first and fourth administration
Esketamine t1/2 - plasma elimination half-life | up to 24 hours following the start of first and fourth administration
Esketamine Tmax - time to reach maximum concentration in plasma | up to 24 hours following the start of first and fourth administration
Esnorketamine AUC0-24h - area under the plasma concentration - time curve from time 0 to 24 h | up to 24 hours following the start of first and fourth administration
Esnorketamine Cmax - maximum plasma concentration | up to 24 hours following the start of first and fourth administration
Esnorketamine Tmax - time to reach maximum concentration in plasma | up to 24 hours following the start of first and fourth administration
Changes between predose and postdose values for each administration in hematology and biochemistry | up to 6 weeks
Changes between predose and postdose values for each administration in vital signs (heart rate, blood pressure, respiratory rate) and urinalysis | up to 8 weeks
Changes between predose and postdose values for each administration in SpO2 (blood oxygen saturation) | up to 2 hours following the start of each administration

CONTACTS AND LOCATIONS:
Locations (12):
- Poland (12):
  - Wojewodzki Szpital im. Jana Pawła II, Bełchatów
  - Wojewodzki Szpital dla Nerwowo i Psychicznie Chorych, Bolesławiec
  - Samodzielny Publiczny Psychiatryczny Zaklad Opieki Zdrowotnej, Choroszcz
  - Szpital Miejski, Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Wojewodzki Szpital dla Nerwowo i Psychicznie Chorych, Gmina Świecie
  - Gornoslaskie Centrum Medyczne, Katowice
  - Specjalistyczny Psychiatryczny Zespol Opieki Zdrowotnej, Lodz
  - Pabianickie Centrum Medyczne, Pabianice
  - Mazowieckie Specalistyczne Centrum Zdrowia, Pruszków
  - Mazowiecki Szpital i Centrum Diagnostyczne Allenort, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw